CLINICAL TRIAL: NCT02755961
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Reducing High-Phosphate Containing Diet Education and Proper Phosphate Binder Intake Education to Serum Phosphate Level Among Maintenance Hemodialysis Patients
Brief Title: Efficacy of Dietary Education and Education on Phosphate Binder Use in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Cheol Jeong, Clinical Assistant Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MED-SUR-15-147
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Hyperphosphatemia; End-stage Renal Disease
Keywords: End-stage renal disease; Phosphate binders; Hyperphosphatemia; Dietary education
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): No intervention was performed
- Education group (Experimental): Dietary education and education on phosphate binder use. Pharmacists instructed patients about how to take phosphate binders properly. Dietitians educated on dietary phosphate restriction.
  Interventions: Behavioral: Dietary education; Behavioral: Education on phosphate binder use

INTERVENTIONS:
Behavioral: Dietary education
  Arms: Education group
Behavioral: Education on phosphate binder use
  Arms: Education group

SUMMARY:
Hyperphosphatemia is an independent risk factor for mortality among dialysis patients. And most phosphate in human is derived from the food. The purpose of this study is to evaluate the efficacy of nutritional consultation and education on phosphate binder among dialysis patients.

DETAILED DESCRIPTION:
Hyperphosphatemia is an independent risk factor for mortality among dialysis patients. Hyperphosphatemia is associated with increased incidence of cardiovascular diseases, and is a mediator to the development of hyperparathyroidism and mineral bone disorder. Phosphate is usually obtained by food intake, and it can be removed by hemodialysis. However, the efficacy of removal is limited, so that dietary education and proper intake of phosphate binder is essential.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease patients whose dialysis vintage is more than 3 months

Exclusion Criteria:

* Patients with liver cirrhosis
* Pregnant patients
* Patients with alimentary tract malabsorption diseases
* History of recent alcohol or drug abuse
* Patients receiving chemotherapy for solid organ tumor
* History of mental illness (major depressive disorder, bipolar disorder, schizophrenia, etc.)
* Patients having difficulty communicating with our medical team (dementia, mental retardation, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who reached Ca x P product lower than 55 | 2-3 month

SECONDARY OUTCOMES:
Changes of MMAS-8 score | 1 month, 2-3 month
Changes of bioequivalent dose of phosphate binder | 2-3 month
Changes of PG-SGA | 2-3 month
Amount of change in dietary phosphorus intake | 2-3 month

CONTACTS AND LOCATIONS:
Overall Officials: Jong Cheol Jeong, MD, Principal Investigator — Clinical Assistant Professor